CLINICAL TRIAL: NCT04160676
Title: The Effect of Hydrocortisone-Ascorbic Acid and Thiamine Therapy on the Outcome of Patients With Sepsis: A Prospective Randomized Double-Blinded Controlled Trial
Brief Title: Therapy With Hydrocortisone, Ascorbic Acid, Thamine in Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mostafa Ismail Sharaf (Unknown); Salah Eldeen Ibrahim Alsherif (Unknown); Mohamed Mohi El deen Abo El yazeed (Unknown)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 33375/09/19
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Sepsis
Keywords: Hydrocortison; Ascorbic acid; Thiamine
MeSH Terms: conditions — Sepsis | interventions — Hydrocortisone; Ascorbic Acid; Thiamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel assignment Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All data will be collected by intensivists who will be blinded about the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): The patients in this group will be managed only according to the surviving sepsis campaign 2016 and the surviving sepsis campaign bundle 2018 update.
  The patients will receive 50 ml normal saline I.V within 30 mins / 6 h, 10 ml normal saline I.V / 6 h, 5 ml normal saline I.V / 12 h.
  Interventions: Drug: Normal saline
- Group II (Experimental): The patients will receive the conventional therapy of sepsis and combined therapy of hydrocortisone (Solucortif® 100 mg , vial, dried powder Pfizer, Egypt) 50 mg diluted in 5 ml normal saline IV / 6 h, ascorbic acid (VITAMIN C-®, Amp, ROTEXMEDICA, Germany, 500mg/5ml) 1.5 gm diluted in 50 ml normal saline IV within 30 min /6 h , and thiamine (Vitamin B1-injektopas®, Ampoule, Germany, 100 mg / 2 ml) 200 mg diluted in 10 ml normal saline IV /12 h This combined therapy will be given for 4 days or to the time of discharge if the admission period is less than 4 days
  Interventions: Drug: Hydrocortisone, Ascorbic acid, Thiamine

INTERVENTIONS:
Drug: Hydrocortisone, Ascorbic acid, Thiamine — Combination of hydrocortisone, ascorbic acid, and thiamine
  Arms: Group II
Drug: Normal saline — Normal saline
  Arms: Group I

SUMMARY:
In this study , we suggest that the use of combination of Hydrocortisone, Ascorbic Acid, and Thiamine in patient with sepsis may decrease mortality rate and improve the outcome.

This study will be carried out at SICU of Tanta University hospitals on Patients aged from 18 to 65 years old who will be presented with sepsis that diagnosed according to the surviving sepsis campaign 2016.

Patients who will meet the previous criteria will be enrolled in the study. The patients will be randomized allocated into two groups by the aid of computer generated software of randomization introduced into sealed closed envelops.

All patients will receive the conventional therapy according to the surviving sepsis campaign 2016 and The Surviving Sepsis Campaign Bundle 2018 Update.

The patients will be allocated randomly into one of the following two groups;-. Group I The patients in this group will be managed only according to the surviving sepsis campaign 2016 and the surviving sepsis campaign bundle 2018 update.

The patients will receive 50 ml normal saline I.V within 30 mins / 6 h, 10 ml normal saline I.V / 6 h, 5 ml normal saline I.V / 12 h.

Group II The patients will receive the conventional therapy of sepsis and combined therapy of hydrocortisone (Solucortif® 100 mg , vial, dried powder Pfizer, Egypt) 50 mg diluted in 5 ml normal saline IV / 6 h, ascorbic acid (VITAMIN C-®, Amp, ROTEXMEDICA, Germany, 500mg/5ml) 1.5 gm diluted in 50 ml normal saline IV within 30 min /6 h , and thiamine (Vitamin B1-injektopas®, Ampoule, Germany, 100 mg / 2 ml) 200 mg diluted in 10 ml normal saline IV /12 h The outcome of the patients, the incidence of organ dysfunction will be assessed.

DETAILED DESCRIPTION:
This prospective randomized controlled double-blinded study will be carried out at surgical intensive care units (SICU) in Tanta University Hospitals for a period of 12 months that may be extended after approval from institutional ethical committee.

An informed written consent will be obtained from the patients or patients' relatives.

They will receive an explanation of the purpose of the study and every patient will have a secret code number.

Research results will be only used for scientific purpose. Any unexpected risk/s appearing during the course of research will be clarified to the participants and to the ethical committee on time, however, the patients that will be enrolled in this study have no expected additional risk as we use Hydrocortisone, Ascorbic acid and Thiamin that have minimal side effects.

*Inclusion criteria: Patients aged from 18 to 65 years old who will be presented with sepsis that diagnosed according to the surviving sepsis campaign 2016(21) and The Surviving Sepsis Campaign Bundle 2018 Update.

*Exclusion Criteria:

* Participant or participants' relatives refusal to continue the study.
* Known or suspected allergy to the studied medications.
* Contraindications to the use of vitamin C as renal stones, Alzheimer's disease and Schizophrenia.
* Pre-existing organ failure or dysfunction not related to the presenting sepsis condition.
* Pregnancy.

Patients who will meet the previous criteria will be enrolled in the study. The patients will be randomized allocated into two groups by the aid of computer generated software of randomization introduced into sealed closed envelops.

All patients will receive the conventional therapy according to the surviving sepsis campaign 2016 and The Surviving Sepsis Campaign Bundle 2018 Update.

An intensivist who has no further role in this research work will help in the preparation of the used medications in syringes that will contain medications in group two and normal saline in group one.

(placebo) -I Group The patients in this group will be managed only according to the surviving sepsis campaign 2016 and the surviving sepsis campaign bundle 2018 update.

The patients will receive 50 ml normal saline I.V within 30 mins / 6 h, 10 ml normal saline I.V / 6 h, 5 ml normal saline I.V / 12 h.

Group II The patients will receive the conventional therapy of sepsis and combined therapy of hydrocortisone (Solucortif® 100 mg , vial, dried powder Pfizer, Egypt) 50 mg diluted in 5 ml normal saline IV / 6 h, ascorbic acid (VITAMIN C-®, Amp, ROTEXMEDICA, Germany, 500mg/5ml) 1.5 gm diluted in 50 ml normal saline IV within 30 min /6 h , and thiamine (Vitamin B1-injektopas®, Ampoule, Germany, 100 mg / 2 ml) 200 mg diluted in 10 ml normal saline IV /12 h This combined therapy will be given for 4 days or to the time of discharge if the admission period is less than 4 days.

*Measurements

All data will be collected by intensivists who will be blinded about the study groups. All the patients will be subjected to the following:

1. Demographic data (age, gender, weight, cause of sepsis).
2. 28th day mortality (If the patient will be discharged, data will be collected by phone calls)
3. Sofa score will be recorded daily and compared during the period of the studied drugs administration.
4. Incidence of organ dysfunction during the period of ICU stay.
5. Mean arterial blood pressure will be recorded every 8 hrs and compared during the period of the studied drugs adminstration.
6. Cardiac index will be measured every 8 hrs using Electrical Cardiometry monitor, ICON Cardiotronics, Inc., La Jolla, CA 92307; Osypka Medical GmbH, Berlin,Germany and will be compared between both groups during the period of the studied drugs adminstration.
7. Total dose of vasopressor therapy.
8. Serum lactate level will be measured daily during the period of the studied drugs administration.
9. Serum pocalcitonin level will be measured at time of starting the studied drugs administration and at the end of it.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 65 years old who will be presented with sepsis that diagnosed according to the surviving sepsis campaign 2016 and The Surviving Sepsis Campaign Bundle 2018 Update

Exclusion Criteria:

* Participant or participants' relatives refusal to continue the study.
* Known or suspected allergy to the studied medications.
* Contraindications to the use of vitamin C as renal stones, Alzheimer's disease and Schizophrenia.
* Pre-existing organ failure or dysfunction not related to the presenting sepsis condition.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
28th day mortality rate. | 28 days
  The incidence of mortality in the first 28 days

SECONDARY OUTCOMES:
Changes in SOFA score | 28 days
  the incidence of organ dysfunction
Changes in serum pocalcitonin level | 7 days
  the plasma level of procalcitonin

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No